CLINICAL TRIAL: NCT00573079
Title: Acute Kidney Injury in Premature Infants
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Kidney Foundation, United States (Other)
Responsible Party: Principal Investigator, David Askenazi, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: X070926014
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Acute Kidney Injury
Keywords: Kidney; Infants
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Premature infants in the NICU; 500-1500g birthweight, >=25 weeks gestation

SUMMARY:
Our first Aim is to describe how common a sudden decrease in renal function happens in premature infants in a neonatal intensive care unit. We also want to see how a sudden loss of renal function affects survival. Finally, we will explore non-invasive markers to identify a sudden decrease in renal function from urinary samples.

DETAILED DESCRIPTION:
Advancements in the field of peri-natal medicine has improved the survival of critically ill neonates but yet many still do not survive, and many more are left with long-term damage to vital organ systems. Very little data is available on the impact that acute kidney injury (AKI) has on survival in premature infants, but adult and pediatric studies that show that even mild AKI independently impacts survival after correcting for severity of illness. The role that AKI impacts survival in premature infants is likely to be greater than adults as this acute injury occurs in context of impaired and ongoing kidney development..

Our ability to improve outcomes in children and adults with AKI has been hampered by the inability to recognize AKI early in the disease process. Thus, the work on early non-invasive biomarkers of renal injury has brought great optimism to the field of AKI. Serum and urinary levels of neutrophil gelatinase-associated lipocalin (NGAL), urinary interleukin 18 (IL-18) others are markedly elevated several hours after AKI as opposed to serum creatinine which takes days to rise after the inciting event. Early non-invasive biomarkers of AKI have not been tested in premature infants.

Inclusion criteria - infants (birthweight 500-1500g) be asked to participate in the study. • Exclusion criteria - Infants with prenatal renal ultrasound diagnosis of severe hydronephrosis or other known renal abnormalities will be excluded

ELIGIBILITY:
Inclusion Criteria:

* 500-1500 grams birthweight
* >=25 weeks gestation

Exclusion Criteria:

* infants who do not survive 24 hours of life
* infants with severe congenital abnormalities

Min Age: 1 Minute | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Premature Infants 500-1500grams birthweight >=25 weeks gestation
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2007-12; Primary Completion 2010-12-31 (Actual); Study Completion 2010-12-31

PRIMARY OUTCOMES:
Characterize the incidence and risk factors in critically ill premature infants | 2 years

SECONDARY OUTCOMES:
Compare hospital of premature infants outcomes with and without AKI. Test ability of known noninvasive urinary biomarkers' ability to detect AKI in premature infants | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- UAB, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Koralkar R, Ambalavanan N, Levitan EB, McGwin G, Goldstein S, Askenazi D. Acute kidney injury reduces survival in very low birth weight infants. Pediatr Res. 2011 Apr;69(4):354-8. doi: 10.1203/PDR.0b013e31820b95ca. PMID 21178824